CLINICAL TRIAL: NCT00948675
Title: A Study of Pemetrexed Plus Carboplatin Followed by Maintenance Pemetrexed vs Paclitaxel Plus Carboplatin and Bevacizumab Followed by Maintenance Bevacizumab in Patients With Advanced NCSLC of Nonsquamous Histology
Brief Title: Study of Participants With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13258; H3E-US-S130 (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2014-04-02 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Advanced Non-Small Cell Lung Cancer
Keywords: Advanced Non-Small Cell Lung Cancer of Nonsquamous Histology; Advanced Lung Cancer; Non-Small Cell Lung Cancer; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Pemetrexed; Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pemetrexed + Carboplatin + Pemetrexed (Experimental): Pemetrexed and Carboplatin followed by Pemetrexed
  Interventions: Drug: Pemetrexed; Drug: Carboplatin
- Paclitaxel + Carboplatin + Bevacizumab (Active Comparator): Paclitaxel, Carboplatin, and Bevacizumab followed by Bevacizumab
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Biological: Bevacizumab

INTERVENTIONS:
Drug: Pemetrexed — Induction therapy: 500 milligrams/square meter (mg/m²) given intravenously every 21 days for 4 cycles. Maintenance therapy: 500 mg/m² given intravenously every 21 days until disease progression or treatment discontinuation.
  Other Names: ALIMTA, LY231514
  Arms: Pemetrexed + Carboplatin + Pemetrexed
Drug: Carboplatin — Induction Therapy (every 21 days for 4 cycles): Area Under the Curve (AUC) 6 [maximum possible dose of 900 milligrams (mg)] intravenously infused over 30 minutes.
Drug: Paclitaxel — Induction Therapy (every 21 days for 4 cycles): 200 mg/m² intravenously infused over 3 hours
  Arms: Paclitaxel + Carboplatin + Bevacizumab
Biological: Bevacizumab — Induction therapy: 15 milligrams/kilogram (mg/kg) given intravenously every 21 days for 4 cycles. Maintenance therapy: 15 mg/kg given intravenously every 21 days until disease progression or treatment discontinuation.
  Arms: Paclitaxel + Carboplatin + Bevacizumab

SUMMARY:
The purpose of this study is to compare the regimens of pemetrexed, carboplatin with pemetrexed maintenance and paclitaxel, carboplatin, bevacizumab with bevacizumab maintenance in participants with Stage IV nonsquamous non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, Phase III trial. Eligible participants will be randomized in a 1:1 ratio to receive pemetrexed and carboplatin followed by pemetrexed or paclitaxel, carboplatin, and bevacizumab followed by bevacizumab as their study treatment. Participants randomized to Pemetrexed + Carboplatin + Pemetrexed will receive folic acid, vitamin B12, and dexamethasone as stated in the pemetrexed label. Before administration of paclitaxel, participants randomized to Paclitaxel + Carboplatin + Bevacizumab will receive premedication (dexamethasone, diphenhydramine, and cimetidine or ranitidine) as recommended in the paclitaxel label.

ELIGIBILITY:
Inclusion Criteria:

* a histologic or cytologic diagnosis of advanced non-small cell lung cancer (NSCLC) [Stage IV from the American Joint Committee on Cancer Staging Criteria (AJCC) staging system, version 7.0, including both M1a and M1b], other than predominantly squamous cell histology, that is not amenable to curative therapy. Participants may not have received any prior systemic chemotherapy, immunotherapy, targeted therapy, or biological therapy, including adjuvant therapy, for any stage of NSCLC.
* prior radiation therapy is allowed to < 25% of the bone marrow; however, prior radiation to the whole pelvis not allowed.
* good performance status.
* adequate organ function.
* estimated life expectancy of at least 12 weeks.

Exclusion Criteria:

* known central nervous system (CNS) disease, other than treated brain metastasis.
* major surgical procedure, open biopsy, open pleurodesis, or significant traumatic injury within 28 days prior to study or have an anticipated need for major surgery during the study.
* core biopsy or other minor surgical procedure, excluding placement of vascular access device, closed pleurodesis, thoracentesis, and mediastinoscopy, within 7 days prior to study.
* history of gastrointestinal fistula, perforation, or abscess, inflammatory bowel disease, or diverticulitis.
* currently receiving ongoing treatment with full-dose warfarin or equivalent
* significant vascular disease within 6 months prior to Day 1 of Cycle 1.
* evidence of bleeding diathesis or coagulopathy.
* serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the participant's ability to adhere to the protocol.
* serious cardiac condition, such as myocardial infarction, angina, or heart disease.
* inadequately controlled hypertension.
* any prior history of hypertensive crisis or hypertensive encephalopathy.
* serious, nonhealing wound, active ulcer, or untreated bone fracture.
* another active malignancy, other than superficial basal cell and superficial squamous (skin) cell, or carcinoma in situ of the cervix within the last 5 years.
* previously received treatment with paclitaxel, carboplatin, pemetrexed, or bevacizumab (prior intravitreal administration of bevacizumab does not preclude study participation).
* pregnant or breast-feeding.
* history of stroke or transient ischemic attack within 6 months prior to study.
* known sensitivity to any component of paclitaxel, carboplatin, pemetrexed, or bevacizumab.
* history of hemoptysis within 3 months prior to randomization.
* unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs).
* unwilling to take folic acid or vitamin B12 supplementation.
* clinically significant third-space fluid collections, for example, ascites or pleural effusions that cannot be controlled by drainage. Participants with M1a disease with pleural effusions are eligible if the effusions can be adequately controlled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2009-09-01 (Actual); Primary Completion 2013-01-31 (Actual); Study Completion 2020-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- United States (45):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scottsdale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mission Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aventura, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gainesville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Port Saint Lucie, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Athens, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Post Falls, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gurnee, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Joliet, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Goshen, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Albany, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mount Sterling, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lansing, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Southfield, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Branson, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Falls, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Burlington, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., High Point, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bismarck, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fargo, North Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tulsa, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DuBois, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nashville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kennewick, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zinner RG, Obasaju CK, Spigel DR, Weaver RW, Beck JT, Waterhouse DM, Modiano MR, Hrinczenko B, Nikolinakos PG, Liu J, Koustenis AG, Winfree KB, Melemed SA, Guba SC, Ortuzar WI, Desaiah D, Treat JA, Govindan R, Ross HJ. PRONOUNCE: randomized, open-label, phase III study of first-line pemetrexed + carboplatin followed by maintenance pemetrexed versus paclitaxel + carboplatin + bevacizumab followed by maintenance bevacizumab in patients ith advanced nonsquamous non-small-cell lung cancer. J Thorac Oncol. 2015 Jan;10(1):134-42. doi: 10.1097/JTO.0000000000000366. PMID 25371077

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who died, participants with progressive disease and those who got randomized but didn't receive any treatment.
Groups:
- Pemetrexed + Carboplatin: Induction therapy: pemetrexed 500 milligrams/square meter (mg/m²) given intravenously plus carboplatin area under the curve (AUC) 6 [maximum possible dose of 900 milligrams (mg)] intravenously infused over 30 minutes for four 21-day cycles.
  Maintenance therapy: pemetrexed 500 mg/m² given intravenously every 21 days until disease progression or treatment discontinuation.
- Paclitaxel + Carboplatin + Bevacizumab: Induction therapy: paclitaxel 200 mg/m² intravenously infused over 3 hours plus carboplatin AUC 6 (maximum possible dose of 900 mg) intravenously infused over 30 minutes plus bevacizumab 15 milligrams/kilogram (mg/kg) given intravenously for four 21-day cycles.
  Maintenance therapy: bevacizumab 15 mg/kg given intravenously every 21 days until disease progression or treatment discontinuation.
Period: Overall Study
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Started | 182 | 179
Received Any Amount of Study Drug | 171 | 166
Completed | 181 | 179
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab | Total
Number analyzed (Participants) | 182 | 179 | 361
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.62) | 64.6 (8.82) | 64.7 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 75 | 152
  Male | 105 | 104 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 178 | 174 | 352
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 20 | 31
  White | 165 | 157 | 322
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 182 | 179 | 361

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Without Grade 4 Toxicity (G4PFS) as Measured by the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Description: G4PFS was defined as the duration from the date of randomization to the earliest occurrence date of one of the following three events: Common Terminology Criteria (CTC) grade 4 adverse events (G4AEs), or progressive disease (PD) or death from any cause, whichever occurred earlier. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PD is ≥20% increase in sum of longest diameter of target lesions or the appearance of new lesions. For participants who had no G4AEs, or PD, or death at the time of the data inclusion cutoff, PFS was censored at their last objective progression-free disease assessment prior to the cutoff date or the date of initiation of subsequent systemic anticancer therapy.
Time Frame: Randomization to measured progressive disease or treatment discontinuation up to 39.49 months
Population: All randomized participants. The number of participants censored was 30 for pemetrexed + carboplatin group and 35 for paclitaxel + carboplatin + bevacizumab group.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Number analyzed (Participants) | 182 | 179
months | 3.91 [2.73 to 4.37] | 2.86 [2.20 to 4.30]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Paclitaxel + Carboplatin + Bevacizumab; Test type: Superiority or Other; p = 0.176, Log Rank

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the duration from the date of randomization to the date of progressive disease (PD) or death from any cause. PD was determined using Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. PD was ≥20% increase in sum of longest diameter of target lesions or the appearance of new lesions. For participants who had no PD or death at the time of the data inclusion cutoff, PFS was censored at their last objective progression-free disease assessment prior to the cutoff date or the date of initiation of subsequent systemic anticancer therapy.
Time Frame: Randomization to measured progressive disease up to 39.49 months
Population: All randomized participants. The number of participants censored was 35 for pemetrexed + carboplatin group and 49 for paclitaxel + carboplatin + bevacizumab group.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Number analyzed (Participants) | 182 | 179
months | 4.44 [4.21 to 5.32] | 5.45 [5.03 to 5.95]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Paclitaxel + Carboplatin + Bevacizumab; Test type: Superiority or Other; p = 0.610, Log Rank

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the duration from the date of randomization to the date of death from any cause. For participants who were alive at the time of the data inclusion cutoff, OS was censored at the last date the participant was known to be alive.
Time Frame: Randomization to date of death from any cause up to 39.49 months
Population: All randomized participants. The number of participants censored was 52 for pemetrexed + carboplatin group and 56 for paclitaxel + carboplatin + bevacizumab group.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Number analyzed (Participants) | 182 | 179
months | 10.51 [9.26 to 11.96] | 11.66 [9.17 to 14.32]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Paclitaxel + Carboplatin + Bevacizumab; Test type: Superiority or Other; p = 0.615, Log Rank

4. Secondary Outcome: Percentage of Participants With Complete Response or Partial Response (Overall Tumor Response Rate)
Description: Overall Response rate (ORR) was the percentage of participants with a confirmed complete response (CR) or partial response (PR), as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR was the disappearance of all target and non-target lesions; PR was a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesions. ORR was calculated as a total number of participants with CR or PR from the start of study treatment until disease progression or recurrence divided by the total number of participants treated, then multiplied by 100.
Time Frame: Baseline to date of objective progressive disease up to 39.49 months
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Number analyzed (Participants) | 182 | 179
percentage of participants | 23.6 [17.7 to 30.5] | 27.4 [21.0 to 34.5]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Paclitaxel + Carboplatin + Bevacizumab; Test type: Superiority or Other; p = 0.414, Pearson Chi-square Test

5. Secondary Outcome: Disease Control Rates Defined as Complete Response (CR), Partial Response (PR), and Stable Disease (SD)
Description: Disease control rate was the percentage of participants with a confirmed CR, PR or SD, as classified by the investigators according to the Response Evaluation Criteria In Solid Tumors (RECIST) criteria version 1.0. CR was the disappearance of all target and non-target lesions; PR was a ≥30% decrease in sum of longest diameter of target lesions without new lesion and progression of non-target lesion; SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Disease control rate was calculated as a total number of participants with CR or PR or SD divided by the total number of participants treated, then multiplied by 100.
Time Frame: Baseline to date of objective progressive disease up to 39.49 months
Population: All randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Number analyzed (Participants) | 182 | 179
percentage of participants | 59.9 [52.4 to 67.1] | 57.0 [49.4 to 64.3]
Statistical Analysis 1: Comparison: Pemetrexed + Carboplatin vs Paclitaxel + Carboplatin + Bevacizumab; Test type: Superiority or Other; p = 0.575, Pearson Chi-square Test

ADVERSE EVENTS:
Time Frame: Baseline to Follow-up (up to 9 years)
Description: Only those participants who received any amount of study drug were included in the safety analysis.
Groups:
- Paclitaxel + Carboplatin + Bevacizumab: Induction therapy: paclitaxel 200 mg/m² intravenously infused over 3 hours plus carboplatin AUC 6 (maximum possible dose of 900 mg) intravenously infused over 30 minutes plus bevacizumab 15 milligrams/kilogram (mg/ kg) given intravenously for four 21-day cycles. Maintenance therapy: bevacizumab 15 mg/kg given intravenously every 21 days until disease progression or treatment discontinuation.
Arm/Group | Pemetrexed + Carboplatin | Paclitaxel + Carboplatin + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 76/171 | 64/166
Other Adverse Events (participants affected / at risk) | 167/171 | 160/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=171) | Paclitaxel + Carboplatin + Bevacizumab (N=166)
Anaemia (Blood and lymphatic system disorders) | 12 (33) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 5 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (8) | 2 (2)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 3 (4) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (3) | 3 (13)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy acute (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (11) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 2 (4) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 6 (12)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Nausea (Gastrointestinal disorders) | 5 (7) | 9 (10)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal obstruction (Gastrointestinal disorders) | 1 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (4) | 10 (12)
Asthenia (General disorders) | 4 (5) | 3 (5)
Catheter site pain (General disorders) | 0 (0) | 1 (2)
Chest pain (General disorders) | 5 (8) | 1 (1)
Disease progression (General disorders) | 3 (4) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 3 (5)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 2 (5) | 1 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (2)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (6)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (15)
Pneumonia (Infections and infestations) | 14 (18) | 6 (13)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 0 (0) | 1 (15)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (4) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 3 (5) | 0 (0)
Platelet count decreased (Investigations) | 2 (3) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 9 (11) | 11 (15)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (7) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (7) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (4)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (4)
Cerebral ischaemia (Nervous system disorders) | 1 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (3)
Embolic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 1 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (5)
Spinal cord compression (Nervous system disorders) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 2 (3)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (3) | 0 (0)
Emotional distress (Psychiatric disorders) | 1 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 3 (4)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (2)
Renal failure (Renal and urinary disorders) | 2 (3) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 4 (4) | 1 (2)
Urinary retention (Renal and urinary disorders) | 1 (2) | 1 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (40) | 2 (8)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (13) | 4 (10)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (10)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 (22) | 5 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 4 (5)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (15) | 3 (3)
Embolism (Vascular disorders) | 0 (0) | 1 (2)
Haematoma (Vascular disorders) | 1 (1) | 1 (2)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 4 (5) | 4 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pemetrexed + Carboplatin (N=171) | Paclitaxel + Carboplatin + Bevacizumab (N=166)
Anaemia (Blood and lymphatic system disorders) | 92 (599) | 59 (380)
Leukopenia (Blood and lymphatic system disorders) | 39 (152) | 32 (89)
Neutropenia (Blood and lymphatic system disorders) | 57 (204) | 80 (270)
Thrombocytopenia (Blood and lymphatic system disorders) | 68 (329) | 47 (154)
Lacrimation increased (Eye disorders) | 14 (107) | 1 (4)
Abdominal pain (Gastrointestinal disorders) | 14 (49) | 14 (29)
Constipation (Gastrointestinal disorders) | 74 (481) | 68 (428)
Diarrhoea (Gastrointestinal disorders) | 30 (108) | 49 (263)
Dyspepsia (Gastrointestinal disorders) | 19 (157) | 15 (75)
Dysphagia (Gastrointestinal disorders) | 4 (25) | 10 (24)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (51) | 10 (121)
Nausea (Gastrointestinal disorders) | 102 (610) | 69 (268)
Stomatitis (Gastrointestinal disorders) | 14 (72) | 15 (46)
Vomiting (Gastrointestinal disorders) | 49 (162) | 32 (83)
Asthenia (General disorders) | 9 (30) | 20 (147)
Chest pain (General disorders) | 17 (62) | 12 (37)
Chills (General disorders) | 12 (21) | 8 (18)
Fatigue (General disorders) | 107 (1045) | 87 (827)
Mucosal inflammation (General disorders) | 11 (39) | 17 (95)
Oedema peripheral (General disorders) | 34 (481) | 12 (71)
Pain (General disorders) | 8 (28) | 9 (64)
Pyrexia (General disorders) | 15 (17) | 11 (15)
Bronchitis (Infections and infestations) | 5 (19) | 12 (21)
Pneumonia (Infections and infestations) | 10 (17) | 6 (20)
Sinusitis (Infections and infestations) | 12 (38) | 12 (31)
Upper respiratory tract infection (Infections and infestations) | 9 (18) | 5 (9)
Urinary tract infection (Infections and infestations) | 20 (34) | 10 (14)
Alanine aminotransferase increased (Investigations) | 14 (58) | 7 (29)
Aspartate aminotransferase increased (Investigations) | 14 (51) | 7 (15)
Blood creatinine increased (Investigations) | 14 (56) | 4 (5)
Haemoglobin decreased (Investigations) | 23 (120) | 8 (51)
Neutrophil count decreased (Investigations) | 12 (43) | 20 (53)
Platelet count decreased (Investigations) | 20 (66) | 8 (43)
Weight decreased (Investigations) | 15 (88) | 30 (155)
White blood cell count decreased (Investigations) | 8 (20) | 12 (25)
Decreased appetite (Metabolism and nutrition disorders) | 52 (281) | 53 (310)
Dehydration (Metabolism and nutrition disorders) | 22 (48) | 20 (66)
Hyperglycaemia (Metabolism and nutrition disorders) | 33 (356) | 22 (104)
Hypokalaemia (Metabolism and nutrition disorders) | 24 (61) | 15 (41)
Hypomagnesaemia (Metabolism and nutrition disorders) | 21 (142) | 24 (86)
Hyponatraemia (Metabolism and nutrition disorders) | 17 (79) | 17 (85)
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 (149) | 38 (285)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (164) | 15 (90)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (38) | 17 (114)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 12 (68) | 6 (19)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (46) | 11 (95)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (70) | 22 (134)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (95) | 19 (88)
Dizziness (Nervous system disorders) | 27 (148) | 20 (64)
Dysgeusia (Nervous system disorders) | 20 (142) | 25 (128)
Headache (Nervous system disorders) | 23 (170) | 25 (213)
Neuropathy peripheral (Nervous system disorders) | 9 (33) | 36 (329)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (83) | 28 (251)
Anxiety (Psychiatric disorders) | 17 (117) | 13 (108)
Depression (Psychiatric disorders) | 12 (160) | 9 (63)
Insomnia (Psychiatric disorders) | 35 (330) | 31 (251)
Proteinuria (Renal and urinary disorders) | 11 (59) | 18 (136)
Cough (Respiratory, thoracic and mediastinal disorders) | 36 (214) | 24 (235)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 (17) | 16 (109)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 (165) | 33 (255)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 17 (49) | 43 (174)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (21) | 10 (19)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (103) | 56 (441)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (112) | 3 (9)
Rash (Skin and subcutaneous tissue disorders) | 21 (83) | 15 (65)
Flushing (Vascular disorders) | 9 (45) | 4 (13)
Hypertension (Vascular disorders) | 3 (12) | 26 (293)
Hypotension (Vascular disorders) | 12 (24) | 11 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days